CLINICAL TRIAL: NCT06502873
Title: Setting up a Cohort of Patients With Inflammatory Bowel Disease and a Cohort of Patients Without Chronic Inflammatory Bowel Disease in the Context of the Translational Study of Biomarkers of Intestinal Dysbiosis (ELITE Walloon Project)
Brief Title: Setting up a Cohort of Patients With Inflammatory Bowel Disease and a Cohort of Patients Without Chronic Inflammatory Bowel Disease
Acronym: ELITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ELITE
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: cohort; BEV; intestinal dysbiosis
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, study aiming to recruit 2 types of patients (60 inflammatory bowel disease (IBD) suffering patients versus 60 control patients without IBD nor any other known intestinal pathology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflammatory bowel disease cohort (Other): 60 patients diagnosed with colonic inflammatory bowel disease
  Interventions: Procedure: biological samples collection
- Control cohort (Other): 60 control patients without inflammatory bowel diseases
  Interventions: Procedure: biological samples collection

INTERVENTIONS:
Procedure: biological samples collection — Collection of biological samples from the same cohorts: faeces, serum, intestinal biopsies

SUMMARY:
The objective of this study is to constitute cohorts of IBD versus non-IBD patients to identify (a) new biomarker(s) of intestinal dysbiosis associated with inflammatory bowel disease, and develop a prototype for assaying such marker(s) in blood.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Male or female ≥ 18 years old
* Able to follow the instructions of the study
* Having signed an informed consent

Specific for Crohn cohort:

* A confirmed diagnosis of IBD
* Rectal or colonic or ileocolic involvement
* Patients with CD presenting inflammatory flare and disease extent in the colon or ileocolic region with:
* A clinical activity defined by an average of four or more instances of very soft or liquid stools daily or an abdominal pain score of 2 or more OR a CDAI (CD Activity Index) ≥ 220 OR a Harvey-Bradshaw Index > 8 OR a faecal calprotectin ≥ 250 µg/g And
* A endoscopic activity defined by a SES-CD (Simple Endoscopic Score for Crohn Disease) ≥ 6 or a CDEIS (CD Endoscopic Index score) ≥ 7
* Patients with UC presenting inflammatory flare with:

A clinical activity defined by a modified Mayo score ≥ 3 OR a Simple Clinical Colitis Activity Index ≥5 OR Patient Reported Outcome (PRO2) ≥ 4 with a subscore of rectal bleeding ≥1 OR a faecal calprotectin ≥ 250 µg/g AND An endoscopic activity defined by a Mayo endoscopic sub-score ≥ 2

Specific for Control cohort:

Patient with no colonic lesion(s) visible during the endoscopical examination (neither Crohn's nor other colitis nor cancer)

Exclusion Criteria:

General criteria:

* Commercial Pharmaceutical probiotic administration within the previous month
* Treatment with antibiotics (whatever the route of administration) within last 3 months
* Non-remission Cancer or in remission for less than 6 months
* Any contraindication to colonoscopy and/or biopsy, left to PI discretion
* Under guardianship or judiciable protection
* Pregnant or breastfeeding women
* Currently participating or having participated in the last 3 months to a clinical study with investigational medicine or food supplement

Specific for Crohn cohort:

* Crohn disease localized only in Ileum
* Inflammatory colon pathology other than Crohn's (infectious, drug-induced,…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited in each cohort | 27 months
  60 patients in IBD cohort and 60 patients in control cohort
number of faeces samples collected in each cohort | 27 months
  60 patients in IBD cohort and 60 patients in control cohort
Number of plasma samples collected in each cohort | 27 months
  60 patients in IBD cohort and 60 patients in control cohort
Number of biopsy samples collected in each cohort | 27 months
  60 patients in IBD cohort and 60 patients in control cohort with 4 colonic biopsies/ patient

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Kemseke, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No